CLINICAL TRIAL: NCT00548262
Title: Open-Label, Non-Comparative, Study Of Intravenous Anidulafungin, Followed Optionally By Oral Voriconazole, For Treatment Of Documented Candidemia/Invasive Candidiasis In Hospitalized Patients
Brief Title: This Is An Open-Label, Non-Comparative Study Designed To Evaluate A Short Course Of IV Anidulafungin, Followed Optionally By Oral Voriconazole, For The Treatment Of Candidemia And Invasive Candidiasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A8851015
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Results first posted 2011-01-17 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2010-12

CONDITIONS: Candidemia; Invasive Candidiasis
Keywords: Open-label; non-comparative study to evaluate short course of IV anidulafungin; followed by oral voriconazole; for tx of candidemia/invasive candidiasis.
MeSH Terms: conditions — Candidemia; Candidiasis, Invasive | interventions — Anidulafungin; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Anidulafungin; Drug: Voriconazole

INTERVENTIONS:
Drug: Anidulafungin — All patients will receive anidulafungin 200 mg IV dose on Day 1. On Day 2 and daily thereafter the patients will receive one daily IV dose of 100 mg of anidulafungin.
  Other Names: Eraxis
Drug: Voriconazole — Patients who complete a minimum of 5 days of IV treatment with anidulafungin may be switched to oral voriconazole 200 mg BID (or 100 mg BID if <40 kg body weight) therapy on Day 5 and thereafter, starting with a loading dose of 400 mg BID (or 200 mg BID if <40 kg body weight).
  Other Names: Vfend

SUMMARY:
The primary objective is to estimate global response rate. Clinical, microbiological and global response rates and its 95% confidence intervals will be computed. No hypotheses will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient 18 years of age and older.
* If female, must be post-menopausal, surgically sterile or using adequate contraception,not lactating, and have a negative urine or blood pregnancy test at screening, prior to administration of study medication.
* Presence of candidemia (positive blood culture) or invasive candidiasis (histopathologic or cytopathologic examination of a needle aspiration or biopsy specimen from a normally sterile site excluding mucous membranes showing yeast cells) obtained within the prior 96 hours to study entry ((informed consent provided).
* Presence of one or more of the following signs and symptoms of acute fungal infection within the prior 48 hours to initiation of study treatment:

  * Fever defined as oral temperature greater than or equal to 38 degrees C (100.4 degrees F); rectal or core temperature greater than or equal to 38.6 degrees C (101.4 degrees F), or axillary temperature greater than or equal to 37.5 degrees Celsius (99.5 degrees F). Hypothermia defined as rectal or core temperature less than 36.0 degrees C (96.8 degrees F).
  * Hypotension (systolic blood pressure [SBP] less than 100 mmHg, or SBP decrease greater than or equal to 30 mm Hg from baseline.
  * Localized signs and symptoms of inflammation (swelling, heat, erythema or purulence at a site infected with Candida spp.).
* Patient is classified in one of following categories based on previous antifungal treatment: received less than 48 hours of previous systemic antifungal therapy and no more than a single dose of echinocandin therapy prior to study entry; intolerant to infusion related toxicities of amphotericin B preparations despite appropriate supportive measures or serum creatinine increased by >1.5 mg/dl while receiving conventional or lipid amphotericin B therapy; or lack of clinical response and/or persistent positive blood culture after at least seven days of systemic antifungal treatment with a polyene or fluconazole at an adequate dose.
* APACHE II 9 score < 25 at study entry.
* Patients willing and able to give informed consent, or have a legally authorized representative willing to give informed consent on the patients behalf.
* Expected survival (in the opinion of the investigator) greater than 4 days.

Exclusion Criteria:

* Hypersensitivity to anidulafungin, other echinocandins or azoles.
* Participation presently or within the last 30 days in a trial with other investigational drug(s). Patients on antiretroviral or chemotherapy regimens which include an investigational drug may participate provided that there has been no change in their therapy during the past 4 weeks and no change in treatment is anticipated during study participation.
* Chronic refractory neutropenia defined as absolute neutrophils count <500 cells/mm3 for 28 days prior to the baseline visit.
* Confirmed or suspected Candida osteomyelitis, endocarditis or meningitis.
* Poor venous access that would preclude IV drug delivery or multiple blood draws.
* Prosthetic devices at a suspected site of infection unless the device is removed within 24 hours of study entry.
* Fungal endophthalmitis confirmed by fundoscopy.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration that may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the Patient inappropriate for entry into this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- Brazil (5):
  - Pfizer Investigational Site, Brasília, Federal District
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São José do Rio Preto, São Paulo
- Pfizer Investigational Site, Independencia, Santiago, RM, Chile
- Colombia (2):
  - Pfizer Investigational Site, Bogota DC, Cundinamarca
  - Pfizer Investigational Site, Cali, Valle del Cauca Department
- Mexico (3):
  - Pfizer Investigational Site, León, Guanajuato
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, San Luis Potosí City, San Luis Potosí
- Pfizer Investigational Site, Panama City, Panama

REFERENCES:
- [Derived] De Rosa FG, Busca A, Capparella MR, Yan JL, Aram JA. Invasive Candidiasis in Patients with Solid Tumors Treated with Anidulafungin: A Post Hoc Analysis of Efficacy and Safety of Six Pooled Studies. Clin Drug Investig. 2021 Jun;41(6):539-548. doi: 10.1007/s40261-021-01024-7. Epub 2021 Apr 23. PMID 33891293
- [Derived] Sganga G, Wang M, Capparella MR, Tawadrous M, Yan JL, Aram JA, Montravers P. Evaluation of anidulafungin in the treatment of intra-abdominal candidiasis: a pooled analysis of patient-level data from 5 prospective studies. Eur J Clin Microbiol Infect Dis. 2019 Oct;38(10):1849-1856. doi: 10.1007/s10096-019-03617-9. Epub 2019 Jul 6. PMID 31280481
- [Derived] Kontoyiannis DP, Bassetti M, Nucci M, Capparella MR, Yan JL, Aram J, Hogan PA. Anidulafungin for the treatment of candidaemia caused by Candida parapsilosis: Analysis of pooled data from six prospective clinical studies. Mycoses. 2017 Oct;60(10):663-667. doi: 10.1111/myc.12641. Epub 2017 Jun 9. PMID 28597967
- [Derived] Kullberg BJ, Vasquez J, Mootsikapun P, Nucci M, Paiva JA, Garbino J, Yan JL, Aram J, Capparella MR, Conte U, Schlamm H, Swanson R, Herbrecht R. Efficacy of anidulafungin in 539 patients with invasive candidiasis: a patient-level pooled analysis of six clinical trials. J Antimicrob Chemother. 2017 Aug 1;72(8):2368-2377. doi: 10.1093/jac/dkx116. PMID 28459966
- [Derived] Nucci M, Colombo AL, Petti M, Magana M, Abreu P, Schlamm HT, Sanchez SP. An open-label study of anidulafungin for the treatment of candidaemia/invasive candidiasis in Latin America. Mycoses. 2014 Jan;57(1):12-8. doi: 10.1111/myc.12094. Epub 2013 May 26. PMID 23710653
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8851015&StudyName=This%20Is%20An%20Open-Label%2C%20Non-Comparative%20Study%20Designed%20To%20Evaluate%20A%20Short%20Course%20Of%20IV%20Anidulafungin%2C%20Followed%20Optionally%20By%20Oral%20Vo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The planned sample size for this study was 210 subjects; however, due to slow enrollment, only 54 subjects were screened and randomized.
Groups:
- Anidulafungin-Voriconazole: Anidulafungin 200 milligrams (mg) intravenously (IV) on Day 1, then once daily 100 mg IV beginning on Day 2. Participants who complete a minimum of 5 days of IV anidulafungin could be switched to oral (PO) voriconazole (loading dose of 400 mg twice daily [BID] or 200 mg BID if body weight < 40 kilograms [kg] and then 200 mg BID or 100 mg BID if body weight < 40 kg thereafter.
Period: Overall Study
Arm/Group | Anidulafungin-Voriconazole
Started | 54 (1 participant (N) had death recorded twice; reported as 1 death in reason for discontinuation (D/C))
Completed | 22 (1 N had D/C recorded as died and as lack of efficacy; reported as lack of efficacy in reason for D/C)
Not Completed | 32
Not completed — Death | 21
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 4
Not completed — Lost to Follow-up | 1
Not completed — Other | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 54
Age, Customized [Number; unit: participants]
  Between 18 and 44 years | 18
  Between 45 and 64 years | 18
  ≥ 65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Global Response (Based on Clinical and Microbiological Success or Failure) at End of Treatment
Description: Clinical Success (cure=resolution of Candida signs and symptoms [s/s] or improvement=significant but incomplete resolution of s/s) or Failure (at least 3 doses Anidulafungin with no significant improvement in s/s or death due to Candida) and Microbiological Success (eradication=negative culture for baseline Candida species (spp) or presumed eradication=follow-up (f/u) culture not available (n/a) and clinical outcome defined as success) or Failure (persistence=positive culture for at least 1 baseline Candida spp or presumed persistence=f/u culture n/a and clinical outcome defined as failure).
Time Frame: End of Treatment (EOT) (up to Day 42)
Population: Modified Intent-to-Treat population (MITT): all Intent-to-Treat (ITT) participants (took at least 1 dose of study treatment) and with a positive baseline culture for a Candida spp within 96 hours before entry into the study. Success=clinical and microbiological success; Failure=all other combinations. Missing or indeterminate set to Failure.
Measure: Number; unit: participants
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 44
participants
  Success | 26 [44.6 to 73.6]
  Failure | 18 [NA to NA]
Statistical Analysis 1: Comparison: Anidulafungin-Voriconazole; Success at EOT; Test type: Superiority or Other; percentage of participants with success = 59.1, 95% CI 2-sided [44.6 to 73.6] — 95% CI based on normal approximation to the binomial

2. Secondary Outcome: Number of Participants for Global Response (Based on Clinical and Microbiological Success or Failure)
Description: as for outcome 1
Time Frame: End of Intravenous Treatment (EIVT) (up to Day 42), Week 2 Follow-up
Population: MITT. Success=clinical and microbiological success; Failure=all other combinations. Missing or indeterminate set to Failure; CI not calculated for Failure.
Measure: Number; unit: participants
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 44
participants
  EIVT Success | 26 [44.6 to 73.6]
  EIVT Failure | 18 [NA to NA]
  Week 2 Follow-up Success | 21 [33.0 to 62.5]
  Week 2 Follow-up Failure | 23 [NA to NA]
Statistical Analysis 1: Comparison: Anidulafungin-Voriconazole; EIVT Success; Test type: Superiority or Other; percentage of participants with success = 59.1, 95% CI 2-sided [44.6 to 73.6] — 95% CI based on normal approximation to the binomial
Statistical Analysis 2: Comparison: Anidulafungin-Voriconazole; Week 2 Follow-up Success; Test type: Superiority or Other; percentage of participants with success = 47.7, 95% CI 2-sided [33.0 to 62.5] — 95% CI based on normal approximation to the binomial

3. Secondary Outcome: Number of Participants for Global Response Per Type of Candida Species Isolated at Baseline: EIVT
Description: Global response based on assessments of Clinical Success or Failure and Microbiological Success or Failure. Categorized as global Success if both clinical and microbiological response=success; Failure defined as all other combinations. Global response at EIVT was assessed per the type of Candida species that was isolated at the baseline visit.
Time Frame: Baseline, EIVT (up to Day 42)
Population: MITT. Missing or indeterminate set to Failure; CI not calculated for Failure.
Measure: Number; unit: participants
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 44
participants
  Candida albicans: Success | 11 [31.0 to 73.7]
  Candida albicans: Failure | 10 [NA to NA]
  Candida famata: Success | 1 [0.0 to 100.0]
  Candida famata: Failure | 1 [NA to NA]
  Candida glabrata: Success | 2 [13.3 to 100.0]
  Candida glabrata: Failure | 1 [NA to NA]
  Candida guilliermondii: Success | 1 [NA to NA]
  Candida guilliermondii: Failure | 0 [NA to NA]
  Candida krusei: Success | 2 [13.3 to 100.0]
  Candida krusei: Failure | 1 [NA to NA]
  Candida parapsilosis: Success | 1 [0.0 to 46.5]
  Candida parapsilosis: Failure | 5 [NA to NA]
  Candida pelliculosa: Success | 1 [NA to NA]
  Candida pelliculosa: Failure | 0 [NA to NA]
  Candida tropicalis: Success | 8 [55.2 to 100.0]
  Candida tropicalis: Failure | 2 [NA to NA]
  Unidentifiable: Success | 4 [20.5 to 93.8]
  Unidentifiable: Failure | 3 [NA to NA]
Statistical Analysis 1: Comparison: Anidulafungin-Voriconazole; Candida albicans: Success; Test type: Superiority or Other; percentage of participants with success = 52.4, 95% CI 2-sided [31.0 to 73.7] — 95% CI based on normal approximation to the binomial
Statistical Analysis 2: Comparison: Anidulafungin-Voriconazole; Candida famata: Success; Test type: Superiority or Other; percentage of participants with success = 50.0, 95% CI 2-sided [0.0 to 100.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 3: Comparison: Anidulafungin-Voriconazole; Candida glabrata: Success; Test type: Superiority or Other; percentage of participants with success = 66.7, 95% CI 2-sided [13.3 to 100.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 4: Comparison: Anidulafungin-Voriconazole; Candida krusei: Success; Test type: Superiority or Other; percentage of participants with success = 66.7, 95% CI 2-sided [13.3 to 100.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 5: Comparison: Anidulafungin-Voriconazole; Candida parapsilosis: Success; Test type: Superiority or Other; percentage of participants with success = 16.7, 95% CI 2-sided [0.0 to 46.5] — 95% CI based on normal approximation to the binomial
Statistical Analysis 6: Comparison: Anidulafungin-Voriconazole; Candida tropicalis: Success; Test type: Superiority or Other; percentage of participants with success = 80.0, 95% CI 2-sided [55.2 to 100.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 7: Comparison: Anidulafungin-Voriconazole; Unidentifiable: Success; Test type: Superiority or Other; percentage of participants with success = 57.1, 95% CI 2-sided [20.5 to 93.8] — 95% CI based on normal approximation to the binomial

4. Secondary Outcome: Number of Participants for Global Response Per Type of Candida Species Isolated at Baseline: EOT
Description: Global response based on assessments of Clinical Success or Failure and Microbiological Success or Failure. Categorized as global Success if both clinical and microbiological response=success; Failure defined as all other combinations. Global response at EOT was assessed per the type of Candida species that was isolated at the baseline visit.
Time Frame: Baseline, EOT (up to Day 42)
Population: MITT. Missing or indeterminate set to Failure; CI not calculated for Failure.
Measure: Number; unit: participants
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 44
participants
  Candida albicans: Success | 11 [31.0 to 73.7]
  Candida albicans: Failure | 10 [NA to NA]
  Candida famata: Success | 0 [NA to NA]
  Candida famata: Failure | 2 [NA to NA]
  Candida glabrata: Success | 2 [13.3 to 100.0]
  Candida glabrata: Failure | 1 [NA to NA]
  Candida guilliermondii: Success | 1 [NA to NA]
  Candida guilliermondii: Failure | 0 [NA to NA]
  Candida krusei: Success | 2 [13.3 to 100.0]
  Candida krusei: Failure | 1 [NA to NA]
  Candida parapsilosis: Success | 1 [0.0 to 46.5]
  Candida parapsilosis: Failure | 5 [NA to NA]
  Candida pelliculosa: Success | 1 [NA to NA]
  Candida pelliculosa: Failure | 0 [NA to NA]
  Candida tropicalis: Success | 8 [55.2 to 100.0]
  Candida tropicalis: Failure | 2 [NA to NA]
  Unidentifiable: Success | 4 [20.5 to 93.8]
  Unidentifiable: Failure | 3 [NA to NA]
Statistical Analysis 1: Comparison: Anidulafungin-Voriconazole; Candida albicans: Success; Test type: Superiority or Other; percentage of participants with success = 52.4, 95% CI 2-sided [31.0 to 73.7] — 95% CI based on normal approximation to the binomial
Statistical Analysis 2: Comparison: Anidulafungin-Voriconazole; Candida glabrata: Success; Test type: Superiority or Other; percentage of participants with success = 66.7, 95% CI 2-sided [13.3 to 100.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 3: Comparison: Anidulafungin-Voriconazole; Candida krusei: Success; Test type: Superiority or Other; percentage of participants with success = 66.7, 95% CI 2-sided [13.3 to 100.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 4: Comparison: Anidulafungin-Voriconazole; Candida parapsilosis: Success; Test type: Superiority or Other; percentage of participants with success = 16.7, 95% CI 2-sided [0.0 to 46.5] — 95% CI based on normal approximation to the binomial
Statistical Analysis 5: Comparison: Anidulafungin-Voriconazole; Candida tropicalis: Success; Test type: Superiority or Other; percentage of participants with success = 80.0, 95% CI 2-sided [55.2 to 100.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 6: Comparison: Anidulafungin-Voriconazole; Unidentifiable: Success; Test type: Superiority or Other; percentage of participants with success = 57.1, 95% CI 2-sided [20.5 to 93.8] — 95% CI based on normal approximation to the binomial

5. Secondary Outcome: Number of Participants for Global Response Per Type of Candida Species Isolated at Baseline: Week 2 Follow-up
Description: Global response based on assessments of Clinical Success or Failure and Microbiological Success or Failure. Categorized as global Success if both clinical and microbiological response=success; Failure defined as all other combinations. Global response at Week 2 Follow-up was assessed per the type of Candida species that was isolated at the baseline visit.
Time Frame: Baseline, Week 2 Follow-up
Population: MITT. Missing or indeterminate set to Failure; CI was not calculated for status of Failure.
Measure: Number; unit: participants
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 44
participants
  Candida albicans: Success | 10 [26.3 to 69.0]
  Candida albicans: Failure | 11 [NA to NA]
  Candida famata: Success | 0 [NA to NA]
  Candida famata: Failure | 2 [NA to NA]
  Candida glabrata: Success | 3 [NA to NA]
  Candida glabrata: Failure | 0 [NA to NA]
  Candida guilliermondii: Success | 1 [NA to NA]
  Candida guilliermondii: Failure | 0 [NA to NA]
  Candida krusei: Success | 2 [13.3 to 100.0]
  Candida krusei: Failure | 1 [NA to NA]
  Candida parapsilosis: Success | 0 [NA to NA]
  Candida parapsilosis: Failure | 6 [NA to NA]
  Candida pelliculosa: Success | 1 [NA to NA]
  Candida pelliculosa: Failure | 0 [NA to NA]
  Candida tropicalis: Success | 7 [41.6 to 98.4]
  Candida tropicalis: Failure | 3 [NA to NA]
  Unidentifiable: Success | 2 [0.0 to 62.0]
  Unidentifiable: Failure | 5 [NA to NA]
Statistical Analysis 1: Comparison: Anidulafungin-Voriconazole; Candida albicans: Success; Test type: Superiority or Other; percentage of participants with success = 47.6, 95% CI 2-sided [26.3 to 69.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 2: Comparison: Anidulafungin-Voriconazole; Candida krusei: Success; Test type: Superiority or Other; percentage of participants with success = 66.7, 95% CI 2-sided [13.3 to 100.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 3: Comparison: Anidulafungin-Voriconazole; Candida tropicalis: Success; Test type: Superiority or Other; percentage of participants with success = 70.0, 95% CI 2-sided [41.6 to 98.4] — 95% CI based on normal approximation to the binomial
Statistical Analysis 4: Comparison: Anidulafungin-Voriconazole; Unidentifiable: Success; Test type: Superiority or Other; percentage of participants with success = 28.6, 95% CI 2-sided [0.0 to 62.0] — 95% CI based on normal approximation to the binomial

6. Secondary Outcome: Number of Participants for Global Response for Pre-specified Baseline Risk Factors Subgroups of Interest: EOT
Description: Global response based on assessments of Clinical Success or Failure and Microbiological Success or Failure. Global response at EOT was assessed for participants categorized with baseline risk factors (Yes or No status) for Intensive Care Unit (ICU) stay ≥ 4 days, mechanical ventilation, broad spectrum antibiotics (antibiotics), central venous (CV) catheter, total parental nutrition (TPN), dialysis, abdominal surgery, solid organ transplant, renal insufficiency, chemotherapy, pancreatitis, systemic steroids or immunosuppressives (Systemic steroids/immunos), neutropenic status, or elderly.
Time Frame: Baseline, EOT (up to Day 42)
Population: MITT. Global Success if both clinical and microbiological response=success; Failure=all other combinations. Missing or indeterminate set to Failure; CI not calculated for failure. Due to small sample size, data was insufficient for analysis by status=elderly (>65 years of age); not summarized.
Measure: Number; unit: participants
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 44
participants
  ICU stay ≥ 4 days (Yes): Success | 18 [39.1 to 73.4]
  ICU stay ≥ 4 days (Yes): Failure | 14 [NA to NA]
  ICU stay ≥ 4 days (No): Success | 8 [40.0 to 93.3]
  ICU stay ≥ 4 days (No): Failure | 4 [NA to NA]
  Mechanical ventilation (Yes): Success | 18 [37.6 to 71.5]
  Mechanical ventilation (Yes): Failure | 15 [NA to NA]
  Mechanical ventilation (No): Success | 8 [46.4 to 99.0]
  Mechanical ventilation (No): Failure | 3 [NA to NA]
  Antibiotics (Yes): Success | 22 [40.8 to 72.0]
  Antibiotics (Yes): Failure | 17 [NA to NA]
  Antibiotics (No): Success | 4 [44.9 to 100.0]
  Antibiotics (No): Failure | 1 [NA to NA]
  CV Catheter (Yes): Success | 21 [39.5 to 71.1]
  CV Catheter (Yes): Failure | 17 [NA to NA]
  CV Catheter (No): Success | 5 [53.5 to 100.0]
  CV Catheter (No): Failure | 1 [NA to NA]
  TPN (Yes): Success | 5 [12.0 to 64.9]
  TPN (Yes): Failure | 8 [NA to NA]
  TPN (No): Success | 21 [51.3 to 84.2]
  TPN (No): Failure | 10 [NA to NA]
  Dialysis (Yes): Success | 3 [6.2 to 79.5]
  Dialysis (Yes): Failure | 4 [NA to NA]
  Dialysis (No): Success | 23 [46.5 to 77.8]
  Dialysis (No): Failure | 14 [NA to NA]
  Abdominal surgery (Yes): Success | 11 [35.7 to 80.1]
  Abdominal surgery (Yes): Failure | 8 [NA to NA]
  Abdominal surgery (No): Success | 15 [40.8 to 79.2]
  Abdominal surgery (No): Failure | 10 [NA to NA]
  Solid organ transplant (No): Success | 26 [44.6 to 73.6]
  Solid organ transplant (No): Failure | 18 [NA to NA]
  Renal insufficiency (Yes): Success | 3 [6.2 to 79.5]
  Renal insufficiency (Yes): Failure | 4 [NA to NA]
  Renal insufficiency (No): Success | 23 [46.5 to 77.8]
  Renal insufficiency (No): Failure | 14 [NA to NA]
  Chemotherapy (Yes): Success | 1 [NA to NA]
  Chemotherapy (Yes): Failure | 0 [NA to NA]
  Chemotherapy (No): Success | 25 [43.4 to 72.9]
  Chemotherapy (No): Failure | 18 [NA to NA]
  Pancreatitis (Yes): Success | 1 [0.0 to 55.1]
  Pancreatitis (Yes): Failure | 4 [NA to NA]
  Pancreatitis (No): Success | 25 [49.0 to 79.2]
  Pancreatitis (No): Failure | 14 [NA to NA]
  Systemic steroids/immunos (Yes): Success | 6 [21.7 to 78.3]
  Systemic steroids/immunos (Yes): Failure | 6 [NA to NA]
  Systemic steroids/immunos (No): Success | 20 [45.7 to 79.3]
  Systemic steroids/immunos (No): Failure | 12 [NA to NA]
  Neutropenic: Success | 2 [13.3 to 100.0]
  Neutropenic: Failure | 1 [NA to NA]
  Non-neutropenic: Success | 18 [44.4 to 79.7]
  Non-neutropenic: Failure | 11 [NA to NA]
Statistical Analysis 1: Comparison: Anidulafungin-Voriconazole; ICU stay ≥ 4 days (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 56.3, 95% CI 2-sided [39.1 to 73.4] — 95% CI based on normal approximation to the binomial
Statistical Analysis 2: Comparison: Anidulafungin-Voriconazole; ICU stay ≥ 4 days (No): Success; Test type: Superiority or Other; percentage of participants with success = 66.7, 95% CI 2-sided [40.0 to 93.3] — 95% CI based on normal approximation to the binomial
Statistical Analysis 3: Comparison: Anidulafungin-Voriconazole; Mechanical ventilation (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 54.5, 95% CI 2-sided [37.6 to 71.5] — 95% CI based on normal approximation to the binomial
Statistical Analysis 4: Comparison: Anidulafungin-Voriconazole; Mechanical ventilation (No): Success; Test type: Superiority or Other; percentage of participants with success = 72.7, 95% CI 2-sided [46.4 to 99.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 5: Comparison: Anidulafungin-Voriconazole; Antibiotics (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 56.4, 95% CI 2-sided [40.8 to 72.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 6: Comparison: Anidulafungin-Voriconazole; Antibiotics (No): Success; Test type: Superiority or Other; percentage of participants with success = 80.0, 95% CI 2-sided [44.9 to 100.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 7: Comparison: Anidulafungin-Voriconazole; CV Catheter (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 55.3, 95% CI 2-sided [39.5 to 71.1] — 95% CI based on normal approximation to the binomial
Statistical Analysis 8: Comparison: Anidulafungin-Voriconazole; CV Catheter (No): Success; Test type: Superiority or Other; percentage of participants with success = 83.3, 95% CI 2-sided [53.5 to 100.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 9: Comparison: Anidulafungin-Voriconazole; TPN (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 38.5, 95% CI 2-sided [12.0 to 64.9] — 95% CI based on normal approximation to the binomial
Statistical Analysis 10: Comparison: Anidulafungin-Voriconazole; TPN (No): Success; Test type: Superiority or Other; percentage of participants with success = 67.7, 95% CI 2-sided [51.3 to 84.2] — 95% CI based on normal approximation to the binomial
Statistical Analysis 11: Comparison: Anidulafungin-Voriconazole; Dialysis (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 42.9, 95% CI 2-sided [6.2 to 79.5] — 95% CI based on normal approximation to the binomial
Statistical Analysis 12: Comparison: Anidulafungin-Voriconazole; Dialysis (No): Success; Test type: Superiority or Other; percentage of participants with success = 62.2, 95% CI 2-sided [46.5 to 77.8] — 95% CI based on normal approximation to the binomial
Statistical Analysis 13: Comparison: Anidulafungin-Voriconazole; Abdominal surgery (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 57.9, 95% CI 2-sided [35.7 to 80.1] — 95% CI based on normal approximation to the binomial
Statistical Analysis 14: Comparison: Anidulafungin-Voriconazole; Abdominal surgery (No): Success; Test type: Superiority or Other; percentage of participants with success = 60.0, 95% CI 2-sided [40.8 to 79.2] — 95% CI based on normal approximation to the binomial
Statistical Analysis 15: Comparison: Anidulafungin-Voriconazole; Solid organ transplant (No): Success; Test type: Superiority or Other; percentage of participants with success = 59.1, 95% CI 2-sided [44.6 to 73.6] — 95% CI based on normal approximation to the binomial
Statistical Analysis 16: Comparison: Anidulafungin-Voriconazole; Renal insufficiency (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 42.9, 95% CI 2-sided [6.2 to 79.5] — 95% CI based on normal approximation to the binomial
Statistical Analysis 17: Comparison: Anidulafungin-Voriconazole; Renal insufficiency (No): Success; Test type: Superiority or Other; percentage of participants with success = 62.2, 95% CI 2-sided [46.5 to 77.8] — 95% CI based on normal approximation to the binomial
Statistical Analysis 18: Comparison: Anidulafungin-Voriconazole; Chemotherapy (No): Success; Test type: Superiority or Other; percentage of participants with success = 58.1, 95% CI 2-sided [43.4 to 72.9] — 95% CI based on normal approximation to the binomial
Statistical Analysis 19: Comparison: Anidulafungin-Voriconazole; Pancreatitis (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 20.0, 95% CI 2-sided [0.0 to 55.1] — 95% CI based on normal approximation to the binomial
Statistical Analysis 20: Comparison: Anidulafungin-Voriconazole; Pancreatitis (No): Success; Test type: Superiority or Other; percentage of participants with success = 64.1, 95% CI 2-sided [49.0 to 79.2] — 95% CI based on normal approximation to the binomial
Statistical Analysis 21: Comparison: Anidulafungin-Voriconazole; Systemic steroids/immunos (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 50.0, 95% CI 2-sided [21.7 to 78.3] — 95% CI based on normal approximation to the binomial
Statistical Analysis 22: Comparison: Anidulafungin-Voriconazole; Systemic steroids/immunos (No): Success; Test type: Superiority or Other; percentage of participants with success = 62.5, 95% CI 2-sided [45.7 to 79.3] — 95% CI based on normal approximation to the binomial
Statistical Analysis 23: Comparison: Anidulafungin-Voriconazole; Neutropenic: Success; Test type: Superiority or Other; percentage of participants with success = 66.7, 95% CI 2-sided [13.3 to 100.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 24: Comparison: Anidulafungin-Voriconazole; Non-neutropenic: Success; Test type: Superiority or Other; percentage of participants with success = 62.1, 95% CI 2-sided [44.4 to 79.7] — 95% CI based on normal approximation to the binomial

7. Secondary Outcome: Number of Participants for Global Response for Baseline Risk Factors for Candidemia and Invasive Candidiasis: EIVT
Description: Global response based on assessments of Clinical Success or Failure and Microbiological Success or Failure. Global response at EIVT was assessed for participants categorized with baseline risk factors for Candidemia and Invasive Candidiasis: ICU stay ≥ 4 days, mechanical ventilation, broad spectrum antibiotics (antibiotics), central venous (CV) catheter, total parental nutrition (TPN), dialysis, abdominal surgery, solid organ transplant, renal insufficiency, chemotherapy, pancreatitis, systemic steroids or immunosuppressives (Systemic steroids/immunos), neutropenic status, or elderly.
Time Frame: EIVT (up to Day 42)
Population: MITT. Global Success if both clinical and microbiological response=success; Failure=all other combinations. Missing or indeterminate set to Failure; CI not calculated for failure. Due to small sample size, data was insufficient for analysis by status=elderly >65 years of age; not summarized.
Measure: Number; unit: participants
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 44
participants
  ICU stay ≥ 4 days (Yes): Success | 18 [39.1 to 73.4]
  ICU stay ≥ 4 days (Yes): Failure | 14 [NA to NA]
  ICU stay ≥ 4 days (No): Success | 8 [40.0 to 93.3]
  ICU stay ≥ 4 days (No): Failure | 4 [NA to NA]
  Mechanical ventilation (Yes): Success | 18 [37.6 to 71.5]
  Mechanical ventilation (Yes): Failure | 15 [NA to NA]
  Mechanical ventilation (No): Success | 8 [46.4 to 99.0]
  Mechanical ventilation (No): Failure | 3 [NA to NA]
  Antibiotics (Yes): Success | 22 [40.8 to 72.0]
  Antibiotics (Yes): Failure | 17 [NA to NA]
  Antibiotics (No): Success | 4 [44.9 to 100.0]
  Antibiotics (No): Failure | 1 [NA to NA]
  CV Catheter (Yes): Success | 21 [39.5 to 71.1]
  CV Catheter (Yes): Failure | 17 [NA to NA]
  CV Catheter (No): Success | 5 [53.5 to 100.0]
  CV Catheter (No): Failure | 1 [NA to NA]
  TPN (Yes): Success | 6 [19.1 to 73.3]
  TPN (Yes): Failure | 7 [NA to NA]
  TPN (No): Success | 20 [47.7 to 81.4]
  TPN (No): Failure | 11 [NA to NA]
  Dialysis (Yes): Success | 3 [6.2 to 79.5]
  Dialysis (Yes): Failure | 4 [NA to NA]
  Dialysis (No): Success | 23 [46.5 to 77.8]
  Dialysis (No): Failure | 14 [NA to NA]
  Abdominal surgery (Yes): Success | 12 [41.5 to 84.8]
  Abdominal surgery (Yes): Failure | 7 [NA to NA]
  Abdominal surgery (No): Success | 14 [36.5 to 75.5]
  Abdominal surgery (No): Failure | 11 [NA to NA]
  Solid organ transplant (No): Success | 26 [44.6 to 73.6]
  Solid organ transplant (No): Failure | 18 [NA to NA]
  Renal insufficiency (Yes): Success | 3 [6.2 to 79.5]
  Renal insufficiency (Yes): Failure | 4 [NA to NA]
  Renal insufficiency (No): Success | 23 [46.5 to 77.8]
  Renal insufficiency (No): Failure | 14 [NA to NA]
  Chemotherapy (Yes): Success | 1 [NA to NA]
  Chemotherapy (Yes): Failure | 0 [NA to NA]
  Chemotherapy (No): Success | 25 [43.4 to 72.9]
  Chemotherapy (No): Failure | 18 [NA to NA]
  Pancreatitis (Yes): Success | 2 [0.0 to 82.9]
  Pancreatitis (Yes): Failure | 3 [NA to NA]
  Pancreatitis (No): Success | 24 [46.3 to 76.8]
  Pancreatitis (No): Failure | 15 [NA to NA]
  Systemic steroids/immunos (Yes): Success | 7 [30.4 to 86.2]
  Systemic steroids/immunos (Yes): Failure | 5 [NA to NA]
  Systemic steroids/immunos (No): Success | 19 [42.4 to 76.4]
  Systemic steroids/immunos (No): Failure | 13 [NA to NA]
  Neutropenic: Success | 2 [13.3 to 100.0]
  Neutropenic: Failure | 1 [NA to NA]
  Non-neutropenic: Success | 18 [44.4 to 79.7]
  Non-neutropenic: Failure | 11 [NA to NA]
Statistical Analysis 1: Comparison: Anidulafungin-Voriconazole; ICU stay ≥ 4 days (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 56.3, 95% CI 2-sided [39.1 to 73.4] — 95% CI based on normal approximation to the binomial
Statistical Analysis 2: Comparison: Anidulafungin-Voriconazole; ICU stay ≥ 4 days (No): Success; Test type: Superiority or Other; percentage of participants with success = 66.7, 95% CI 2-sided [40.0 to 93.3] — 95% CI based on normal approximation to the binomial
Statistical Analysis 3: Comparison: Anidulafungin-Voriconazole; Mechanical ventilation (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 54.5, 95% CI 2-sided [37.6 to 71.5] — 95% CI based on normal approximation to the binomial
Statistical Analysis 4: Comparison: Anidulafungin-Voriconazole; Mechanical ventilation (No): Success; Test type: Superiority or Other; percentage of participants with success = 72.7, 95% CI 2-sided [46.4 to 99.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 5: Comparison: Anidulafungin-Voriconazole; Antibiotics (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 56.4, 95% CI 2-sided [40.8 to 72.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 6: Comparison: Anidulafungin-Voriconazole; Antibiotics (No): Success; Test type: Superiority or Other; percentage of participants with success = 80.0, 95% CI 2-sided [44.9 to 100.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 7: Comparison: Anidulafungin-Voriconazole; CV Catheter (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 55.3, 95% CI 2-sided [39.5 to 71.1] — 95% CI based on normal approximation to the binomial
Statistical Analysis 8: Comparison: Anidulafungin-Voriconazole; CV Catheter (No): Success; Test type: Superiority or Other; percentage of participants with success = 83.3, 95% CI 2-sided [53.5 to 100.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 9: Comparison: Anidulafungin-Voriconazole; TPN (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 46.2, 95% CI 2-sided [19.1 to 73.3] — 95% CI based on normal approximation to the binomial
Statistical Analysis 10: Comparison: Anidulafungin-Voriconazole; TPN (No): Success; Test type: Superiority or Other; percentage of participants with success = 64.5, 95% CI 2-sided [47.7 to 81.4] — 95% CI based on normal approximation to the binomial
Statistical Analysis 11: Comparison: Anidulafungin-Voriconazole; Dialysis (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 42.9, 95% CI 2-sided [6.2 to 79.5] — 95% CI based on normal approximation to the binomial
Statistical Analysis 12: Comparison: Anidulafungin-Voriconazole; Dialysis (No): Success; Test type: Superiority or Other; percentage of participants with success = 62.2, 95% CI 2-sided [46.5 to 77.8] — 95% CI based on normal approximation to the binomial
Statistical Analysis 13: Comparison: Anidulafungin-Voriconazole; Abdominal surgery (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 63.2, 95% CI 2-sided [41.5 to 84.8] — 95% CI based on normal approximation to the binomial
Statistical Analysis 14: Comparison: Anidulafungin-Voriconazole; Abdominal surgery (No): Success; Test type: Superiority or Other; percentage of participants with success = 56.0, 95% CI 2-sided [36.5 to 75.5] — 95% CI based on normal approximation to the binomial
Statistical Analysis 15: Comparison: Anidulafungin-Voriconazole; Solid organ transplant (No): Success; Test type: Superiority or Other; percentage of participants with success = 59.1, 95% CI 2-sided [44.6 to 73.6] — 95% CI based on normal approximation to the binomial
Statistical Analysis 16: Comparison: Anidulafungin-Voriconazole; Renal insufficiency (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 42.9, 95% CI 2-sided [6.2 to 79.5] — 95% CI based on normal approximation to the binomial
Statistical Analysis 17: Comparison: Anidulafungin-Voriconazole; Renal insufficiency (No): Success; Test type: Superiority or Other; percentage of participants with success = 62.2, 95% CI 2-sided [46.5 to 77.8] — 95% CI based on normal approximation to the binomial
Statistical Analysis 18: Comparison: Anidulafungin-Voriconazole; Chemotherapy (No): Success; Test type: Superiority or Other; percentage of participants with success = 58.1, 95% CI 2-sided [43.4 to 72.9] — 95% CI based on normal approximation to the binomial
Statistical Analysis 19: Comparison: Anidulafungin-Voriconazole; Pancreatitis (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 40.0, 95% CI 2-sided [0.0 to 82.9] — 95% CI based on normal approximation to the binomial
Statistical Analysis 20: Comparison: Anidulafungin-Voriconazole; Pancreatitis (No): Success; Test type: Superiority or Other; percentage of participants with success = 61.5, 95% CI 2-sided [46.3 to 76.8] — 95% CI based on normal approximation to the binomial
Statistical Analysis 21: Comparison: Anidulafungin-Voriconazole; Systemic steroids/immunos (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 58.3, 95% CI 2-sided [30.4 to 86.2] — 95% CI based on normal approximation to the binomial
Statistical Analysis 22: Comparison: Anidulafungin-Voriconazole; Systemic steroids/immunos (No): Success; Test type: Superiority or Other; percentage of participants with success = 59.4, 95% CI 2-sided [42.4 to 76.4] — 95% CI based on normal approximation to the binomial
Statistical Analysis 23: Comparison: Anidulafungin-Voriconazole; Neutropenic: Success; Test type: Superiority or Other; percentage of participants with success = 66.7, 95% CI 2-sided [13.3 to 100.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 24: Comparison: Anidulafungin-Voriconazole; Non-neutropenic: Success; Test type: Superiority or Other; percentage of participants with success = 62.1, 95% CI 2-sided [44.4 to 79.7] — 95% CI based on normal approximation to the binomial

8. Secondary Outcome: Number of Participants for Global Response for Baseline Risk Factors for Candidemia and Invasive Candidiasis: Week 2 Follow-up
Description: Global response based on assessments of Clinical Success or Failure and Microbiological Success or Failure. Global response at Week 2 F/U was assessed for participants categorized with baseline risk factors for Candidemia and Invasive Candidiasis: ICU stay ≥ 4 days, mechanical ventilation, broad spectrum antibiotics (antibiotics), central venous (CV) catheter, total parental nutrition (TPN), dialysis, abdominal surgery, solid organ transplant, renal insufficiency, chemotherapy, pancreatitis, systemic steroids or immunosuppressives (Systemic steroids/immunos), neutropenic status, or elderly.
Time Frame: Baseline, Week 2 Follow-up (F/U)
Population: MITT. Global Success if both clinical and microbiological response=success; Failure=all other combinations. Missing or indeterminate set to Failure; CI not calculated for failure. Due to small sample size, data insufficient for analysis by status=elderly >65 years of age; not summarized.
Measure: Number; unit: participants
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 44
participants
  ICU stay ≥ 4 days (Yes): Success | 12 [20.7 to 54.3]
  ICU stay ≥ 4 days (Yes): Failure | 20 [NA to NA]
  ICU stay ≥ 4 days (No): Success | 9 [50.5 to 99.5]
  ICU stay ≥ 4 days (No): Failure | 3 [NA to NA]
  Mechanical ventilation (Yes): Success | 13 [22.7 to 56.1]
  Mechanical ventilation (Yes): Failure | 20 [NA to NA]
  Mechanical ventilation (No): Success | 8 [46.4 to 99.0]
  Mechanical ventilation (No): Failure | 3 [NA to NA]
  Antibiotics (Yes): Success | 19 [33.0 to 64.4]
  Antibiotics (Yes): Failure | 20 [NA to NA]
  Antibiotics (No): Success | 2 [0.0 to 82.9]
  Antibiotics (No): Failure | 3 [NA to NA]
  CV Catheter (Yes): Success | 18 [31.5 to 63.2]
  CV Catheter (Yes): Failure | 20 [NA to NA]
  CV Catheter (No): Success | 3 [10.0 to 90.0]
  CV Catheter (No): Failure | 3 [NA to NA]
  TPN (Yes): Success | 5 [12.0 to 64.9]
  TPN (Yes): Failure | 8 [NA to NA]
  TPN (No): Success | 16 [34.0 to 69.2]
  TPN (No): Failure | 15 [NA to NA]
  Dialysis (Yes): Success | 1 [0.0 to 40.2]
  Dialysis (Yes): Failure | 6 [NA to NA]
  Dialysis (No): Success | 20 [38.0 to 70.1]
  Dialysis (No): Failure | 17 [NA to NA]
  Abdominal surgery (Yes): Success | 8 [19.9 to 64.3]
  Abdominal surgery (Yes): Failure | 11 [NA to NA]
  Abdominal surgery (No): Success | 13 [32.4 to 71.6]
  Abdominal surgery (No): Failure | 12 [NA to NA]
  Solid organ transplant (No): Success | 21 [33.0 to 62.5]
  Solid organ transplant (No): Failure | 23 [NA to NA]
  Renal insufficiency (Yes): Success | 1 [0.0 to 40.2]
  Renal insufficiency (Yes): Failure | 6 [NA to NA]
  Renal insufficiency (No): Success | 20 [38.0 to 70.1]
  Renal insufficiency (No): Failure | 17 [NA to NA]
  Chemotherapy (Yes): Success | 1 [NA to NA]
  Chemotherapy (Yes): Failure | 0 [NA to NA]
  Chemotherapy (No): Success | 20 [31.6 to 61.4]
  Chemotherapy (No): Failure | 23 [NA to NA]
  Pancreatitis (Yes): Success | 2 [0.0 to 82.9]
  Pancreatitis (Yes): Failure | 3 [NA to NA]
  Pancreatitis (No): Success | 19 [33.0 to 64.4]
  Pancreatitis (No): Failure | 20 [NA to NA]
  Systemic steroids/immunos (Yes): Success | 5 [13.8 to 69.6]
  Systemic steroids/immunos (Yes): Failure | 7 [NA to NA]
  Systemic steroids/immunos (No): Success | 16 [32.7 to 67.3]
  Systemic steroids/immunos (No): Failure | 16 [NA to NA]
  Neutropenic: Success | 2 [13.3 to 100.0]
  Neutropenic: Failure | 1 [NA to NA]
  Non-neutropenic: Success | 15 [33.5 to 69.9]
  Non-neutropenic: Failure | 14 [NA to NA]
Statistical Analysis 1: Comparison: Anidulafungin-Voriconazole; ICU stay ≥ 4 days (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 37.5, 95% CI 2-sided [20.7 to 54.3] — 95% CI based on normal approximation to the binomial
Statistical Analysis 2: Comparison: Anidulafungin-Voriconazole; ICU stay ≥ 4 days (No): Success; Test type: Superiority or Other; percentage of participants with success = 75.0, 95% CI 2-sided [50.5 to 99.5] — 95% CI based on normal approximation to the binomial
Statistical Analysis 3: Comparison: Anidulafungin-Voriconazole; Mechanical ventilation (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 39.4, 95% CI 2-sided [22.7 to 56.1] — 95% CI based on normal approximation to the binomial
Statistical Analysis 4: Comparison: Anidulafungin-Voriconazole; Mechanical ventilation (No): Success; Test type: Superiority or Other; percentage of participants with success = 72.7, 95% CI 2-sided [46.4 to 99.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 5: Comparison: Anidulafungin-Voriconazole; Antibiotics (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 48.7, 95% CI 2-sided [33.0 to 64.4] — 95% CI based on normal approximation to the binomial
Statistical Analysis 6: Comparison: Anidulafungin-Voriconazole; Antibiotics (No): Success; Test type: Superiority or Other; percentage of participants with success = 40.0, 95% CI 2-sided [0.0 to 82.9] — 95% CI based on normal approximation to the binomial
Statistical Analysis 7: Comparison: Anidulafungin-Voriconazole; CV Catheter (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 47.4, 95% CI 2-sided [31.5 to 63.2] — 95% CI based on normal approximation to the binomial
Statistical Analysis 8: Comparison: Anidulafungin-Voriconazole; CV Catheter (No): Success; Test type: Superiority or Other; percentage of participants with success = 50.0, 95% CI 2-sided [10.0 to 90.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 9: Comparison: Anidulafungin-Voriconazole; TPN (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 38.5, 95% CI 2-sided [12.0 to 64.9] — 95% CI based on normal approximation to the binomial
Statistical Analysis 10: Comparison: Anidulafungin-Voriconazole; TPN (No): Success; Test type: Superiority or Other; percentage of participants with success = 51.6, 95% CI 2-sided [34.0 to 69.2] — 95% CI based on normal approximation to the binomial
Statistical Analysis 11: Comparison: Anidulafungin-Voriconazole; Dialysis (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 14.3, 95% CI 2-sided [0.0 to 40.2] — 95% CI based on normal approximation to the binomial
Statistical Analysis 12: Comparison: Anidulafungin-Voriconazole; Dialysis (No): Success; Test type: Superiority or Other; percentage of participants with success = 54.1, 95% CI 2-sided [38.0 to 70.1] — 95% CI based on normal approximation to the binomial
Statistical Analysis 13: Comparison: Anidulafungin-Voriconazole; Abdominal surgery (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 42.1, 95% CI 2-sided [19.9 to 64.3] — 95% CI based on normal approximation to the binomial
Statistical Analysis 14: Comparison: Anidulafungin-Voriconazole; Abdominal surgery (No): Success; Test type: Superiority or Other; percentage of participants with success = 52.0, 95% CI 2-sided [32.4 to 71.6] — 95% CI based on normal approximation to the binomial
Statistical Analysis 15: Comparison: Anidulafungin-Voriconazole; Solid organ transplant (No): Success; Test type: Superiority or Other; percentage of participants with success = 47.7, 95% CI 2-sided [33.0 to 62.5] — 95% CI based on normal approximation to the binomial
Statistical Analysis 16: Comparison: Anidulafungin-Voriconazole; Renal insufficiency (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 14.3, 95% CI 2-sided [0.0 to 40.2] — 95% CI based on normal approximation to the binomial
Statistical Analysis 17: Comparison: Anidulafungin-Voriconazole; Renal insufficiency (No): Success; Test type: Superiority or Other; percentage of participants with success = 54.1, 95% CI 2-sided [38.0 to 70.1] — 95% CI based on normal approximation to the binomial
Statistical Analysis 18: Comparison: Anidulafungin-Voriconazole; Chemotherapy (No): Success; Test type: Superiority or Other; percentage of participants with success = 46.5, 95% CI 2-sided [31.6 to 61.4] — 95% CI based on normal approximation to the binomial
Statistical Analysis 19: Comparison: Anidulafungin-Voriconazole; Pancreatitis (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 40.0, 95% CI 2-sided [0.0 to 82.9] — 95% CI based on normal approximation to the binomial
Statistical Analysis 20: Comparison: Anidulafungin-Voriconazole; Pancreatitis (No): Success; Test type: Superiority or Other; percentage of participants with success = 48.7, 95% CI 2-sided [33.0 to 64.4] — 95% CI based on normal approximation to the binomial
Statistical Analysis 21: Comparison: Anidulafungin-Voriconazole; Systemic steroids/immunos (Yes): Success; Test type: Superiority or Other; percentage of participants with success = 41.7, 95% CI 2-sided [13.8 to 69.6] — 95% CI based on normal approximation to the binomial
Statistical Analysis 22: Comparison: Anidulafungin-Voriconazole; Systemic steroids/immunos (No): Success; Test type: Superiority or Other; percentage of participants with success = 50.0, 95% CI 2-sided [32.7 to 67.3] — 95% CI based on normal approximation to the binomial
Statistical Analysis 23: Comparison: Anidulafungin-Voriconazole; Neutropenic: Success; Test type: Superiority or Other; percentage of participants with success = 66.7, 95% CI 2-sided [13.3 to 100.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 24: Comparison: Anidulafungin-Voriconazole; Non-neutropenic: Success; Test type: Superiority or Other; percentage of participants with success = 51.7, 95% CI 2-sided [33.5 to 69.9] — 95% CI based on normal approximation to the binomial

9. Secondary Outcome: Number of Participants for Global Response by Acute Physiological Assessment and Chronic Health Evaluation II (APACHE II) Score
Description: Global response based on assessments of Clinical Success or Failure and Microbiological Success or Failure. Categorized as global Success if both clinical and microbiological response=success; Failure defined as all other combinations. Global response assessed as APACHE II score <20 (less affected) or ≥20 (more severe). APACHE II assesses severity of illness in acutely ill participants; measurements computed for physiologic variables were transformed to integer score ranging 0 (normal) to 71 (more severe). Higher scores indicate more severe disease and higher risk of death.
Time Frame: EIVT (up to Day 42), EOT (up to Day 42), Week 2 Follow-up
Population: MITT. Missing or indeterminate set to Failure; CI not calculated for Failure.
Measure: Number; unit: participants
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 44
participants
  APACHE <20 (EIVT): Success | 24 [53.2 to 84.0]
  APACHE <20 (EIVT): Failure | 11 [NA to NA]
  APACHE ≥20 (EIVT): Success | 2 [0.0 to 49.4]
  APACHE ≥20 (EIVT): Failure | 7 [NA to NA]
  APACHE <20 (EOT): Success | 25 [56.5 to 86.4]
  APACHE <20 (EOT): Failure | 10 [NA to NA]
  APACHE ≥20 (EOT): Success | 1 [0.0 to 31.6]
  APACHE ≥20 (EOT): Failure | 8 [NA to NA]
  APACHE <20 (Week 2 F/U): Success | 20 [40.7 to 73.5]
  APACHE <20 (Week 2 F/U): Failure | 15 [NA to NA]
  APACHE ≥20 (Week 2 F/U): Success | 1 [0.0 to 31.6]
  APACHE ≥20 (Week 2 F/U): Failure | 8 [NA to NA]
Statistical Analysis 1: Comparison: Anidulafungin-Voriconazole; APACHE <20 (EIVT): Success; Test type: Superiority or Other; percentage of participants with success = 68.6, 95% CI 2-sided [53.2 to 84.0] — 95% CI based on normal approximation to the binomial
Statistical Analysis 2: Comparison: Anidulafungin-Voriconazole; APACHE ≥20 (EIVT): Success; Test type: Superiority or Other; percentage of participants with success = 22.2, 95% CI 2-sided [0.0 to 49.4] — 95% CI based on normal approximation to the binomial
Statistical Analysis 3: Comparison: Anidulafungin-Voriconazole; APACHE <20 (EOT): Success; Test type: Superiority or Other; percentage of participants with success = 71.4, 95% CI 2-sided [56.5 to 86.4] — 95% CI based on normal approximation to the binomial
Statistical Analysis 4: Comparison: Anidulafungin-Voriconazole; APACHE ≥20 (EOT): Success; Test type: Superiority or Other; percentage of participants with success = 11.1, 95% CI 2-sided [0.0 to 31.6] — 95% CI based on normal approximation to the binomial
Statistical Analysis 5: Comparison: Anidulafungin-Voriconazole; APACHE <20 (Week 2 F/U): Success; Test type: Superiority or Other; percentage of participants with success = 57.1, 95% CI 2-sided [40.7 to 73.5] — 95% CI based on normal approximation to the binomial
Statistical Analysis 6: Comparison: Anidulafungin-Voriconazole; APACHE ≥20 (Week 2 F/U): Success; Test type: Superiority or Other; percentage of participants with success = 11.1, 95% CI 2-sided [0.0 to 31.6] — 95% CI based on normal approximation to the binomial

10. Secondary Outcome: Number of Participants Per Survival Status (Alive or Dead) on Day 30
Time Frame: Day 30
Population: MITT
Measure: Number; unit: participants
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 44
participants
  Alive | 25
  Dead | 19

11. Secondary Outcome: Number of Participants With Death Attributable (Yes or No) to Candidemia or Invasive Candidiasis
Description: Death is attributable to Candidemia or Invasive Candidiasis if investigator recorded "disease under study" as cause of death. Candidemia (positive blood culture) or Invasive Cadidiasis (yeast cells in histopathological or cytopathological exam). Week 6 Follow-up visit conducted by phone.
Time Frame: Baseline to Week 6 Follow-up
Population: MITT. MITT. Death for 1 participant reported twice in this study(recorded at End of Treatment and at End of Study); both instances are reported in this table under Attributal Death=No.
Measure: Number; unit: participants
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 44
participants
  Attributable death (Yes) | 4
  Attributable death (No) | 19

12. Secondary Outcome: Time to Negative Blood, Specimen, or Tissue Culture
Description: Defined as time from first drug administratin to date of earliest recorded documentation of negative blood, specimen, or tissue culture (absence of Candidemia or Invasive Candidiasis). Candidemia (positive blood culture) or Invasive Cadidiasis (yeast cells in histopathological or cytopathological exam).
Time Frame: Baseline to Week 2 Follow-up
Population: MITT; data not summarized using descriptive statistics.
Measure: Number; unit: Days
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 0

13. Secondary Outcome: Duration of Exposure to Intravenous Anidulafungin Prior to Switch to Oral Voriconazole Treatment
Description: Defined as time in days from first intravenous administration of Anidulafungin to the date of earliest recorded documentation of switch to oral Voriconazole treatment. Participants received at least 5 days (and a maximum of 42 days) of IV Anidulafungin; after this, they may continue treatment with oral Voriconazole for at least 14 days from the day of last positive culture up to a maximum of 42 days.
Time Frame: Baseline to Day 42
Population: Safety analysis set: all participants who received any dose of study medication.
Measure: Median (Full Range); unit: days
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 54
days | 10.0 [1 to 28]

14. Secondary Outcome: Length of Hospital Stay
Description: Defined as the number of days from date of first drug administration to date of first hospital discharge if participant was discharged to home or other location. Week 6 Follow-up visit conducted by phone.
Time Frame: Baseline to Week 6 Follow-up
Population: MITT; data not summarized using descriptive statistics.
Measure: Number; unit: days
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 0

15. Secondary Outcome: Length of Stay in Intensive Care Unit (ICU)
Description: Defined as the number of days from date of first drug administration to date of first ICU discharge. Week 6 Follow-up visit conducted by phone.
Time Frame: Baseline up to Week 6 Follow-up
Population: MITT; N=number of participants evaluable for length of time in ICU.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 32
Days | 16.0 [8.0 to 29.0]

16. Secondary Outcome: Change From Baseline in Vital Signs: Supine Blood Pressure
Description: Supine systolic and diastolic blood pressure BP) measured as millimeters of mercury (mmHg).
Time Frame: Baseline to Week 2 Follow-up
Population: Safety analysis population
Measure: Median (Full Range); unit: mmHg
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 54
mmHg
  Baseline median: supine systolic BP | 120.0 [NA to NA] — Measure of dispersion was not calculated for baseline median.
  Change from baseline: supine systolic BP | 0.00 [NA to NA] — Measure of dispersion was not calculated for median change from baseline.
  Baseline median: supine diastolic BP | 66.0 [NA to NA] — Measure of dispersion was not calculated for baseline median.
  Change from baseline: supine diastolic BP | 0.00 [NA to NA] — Measure of dispersion was not calculated for median change from baseline.

17. Secondary Outcome: Change From Baseline in Vital Signs: Supine Heart Rate
Description: Supine heart rate measured as beats per minute (bpm).
Time Frame: Baseline to Week 2 Follow-up
Population: Safety analysis population
Measure: Median (Full Range); unit: bpm
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 54
bpm
  Baseline median: supine heart rate | 97.5 [NA to NA] — Measure of dispersion was not calculated for baseline median.
  Change from baseline: supine heart rate | 3.00 [NA to NA] — Measure of dispersion was not calculated for median change from baseline.

18. Secondary Outcome: Change From Baseline in Vital Signs: Weight
Description: Weight measured as kilograms (kg).
Time Frame: Baseline to Week 2 Follow-up
Population: Safety analysis population; N=number of participants with evaluable data.
Measure: Median (Full Range); unit: kg
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 30
kg
  Baseline median: weight | 65.0 [NA to NA] — Measure of dispersion was not calculated for baseline median.
  Change from baseline: weight | -0.70 [NA to NA] — Measure of dispersion was not calculated for median change from baseline.

19. Secondary Outcome: Change From Baseline in Vital Signs: Temperature
Description: Temperature measured as degrees of Celsius (C).
Time Frame: Baseline to Week 2 Follow-up
Population: Safety analysis population
Measure: Median (Full Range); unit: Degrees of Celsius
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 54
Degrees of Celsius
  Baseline median: temperature | 37.5 [NA to NA] — Measure of dispersion was not calculated for baseline median.
  Change from baseline: temperature | -0.30 [NA to NA] — Measure of dispersion was not calculated for median change from baseline.

20. Secondary Outcome: Change From Baseline in Vital Signs: Respiration Rate
Description: Respiration rate measured as respirations per minute (resp/min).
Time Frame: Baseline to Week 2 Follow-up
Population: Safety analysis population
Measure: Median (Full Range); unit: resp/min
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 54
resp/min
  Baseline median: respiration rate | 20.0 [NA to NA] — Measure of dispersion was not calculated for baseline median.
  Change from baseline: respiration rate | -0.50 [NA to NA] — Measure of dispersion was not calculated for median change from baseline.

21. Secondary Outcome: Change From Baseline in Chemistry Laboratory Test Data (Measured as mg/dL)
Description: Chemistry laboratory test data measured as milligrams per deciliter (mg/dL).
Time Frame: Baseline to Week 2 Follow-up
Population: Safety analysis population; N=number of participants with analyzable laboratory data; (n)=number of subjects with data for each test at observation.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 27
mg/dL
  Baseline median: total bilirubin (n=19) | 0.6 [NA to NA] — Measure of dispersion was not calculated for baseline median.
  Change from baseline: total bilirubin | -0.2 [NA to NA] — Measure of dispersion was not calculated for median change from baseline.
  Baseline median: direct bilirubin (n=19) | 0.2 [NA to NA] — Measure of dispersion was not calculated for baseline median.
  Change from baseline: direct bilirubin | -0.1 [NA to NA] — Measure of dispersion was not calculated for median change from baseline.
  Baseline median: indirect bilirubin (n=17) | 0.3 [NA to NA] — Measure of dispersion was not calculated for baseline median.
  Change from baseline: indirect bilirubin | 0.0 [NA to NA] — Measure of dispersion was not calculated for median change from baseline.
  Baseline median: blood urea nitrogen (n=25) | 37.4 [NA to NA] — Measure of dispersion was not calculated for baseline median.
  Change from baseline: blood urea nitrogen | -4.8 [NA to NA] — Measure of dispersion was not calculated for median change from baseline.
  Baseline median: creatinine (n=27) | 0.8 [NA to NA] — Measure of dispersion was not calculated for baseline median.
  Change from baseline: creatinine | 0.0 [NA to NA] — Measure of dispersion was not calculated for median change from baseline.
  Baseline median: glucose (n=24) | 99 [NA to NA] — Measure of dispersion was not calculated for baseline median.
  Change from baseline: glucose | -6 [NA to NA] — Measure of dispersion was not calculated for median change from baseline.

22. Secondary Outcome: Change From Baseline in Chemistry Laboratory Test Data (Measured as IU/L)
Description: Chemistry laboratory test data measured as international units per (IU/L).
Time Frame: Baseline to Week 2 Follow-up
Population: as for outcome 21
Measure: Median (Full Range); unit: IU/L
Arm/Group | Anidulafungin-Voriconazole
Number analyzed (Participants) | 18
IU/L
  Baseline median: aspartate aminotransferase (n=18) | 43 [NA to NA] — Measure of dispersion was not calculated for baseline median.
  Change from baseline: aspartate aminotransferase | -18 [NA to NA] — Measure of dispersion was not calculated for median change from baseline.
  Baseline median: alanine aminotransferase (n=16) | 45 [NA to NA] — Measure of dispersion was not calculated for baseline median.
  Change from baseline: alanine aminotransferase | -5 [NA to NA] — Measure of dispersion was not calculated for median change from baseline.
  Baseline median: lactate dehydrogenase (n=13) | 536 [NA to NA] — Measure of dispersion was not calculated for baseline median.
  Change from baseline: lactate dehydrogenase | -160 [NA to NA] — Measure of dispersion was not calculated for median change from baseline.
  Baseline median: alkaline phosphatase (n=17) | 114 [NA to NA] — Measure of dispersion was not calculated for baseline median.
  Change from baseline: alkaline phosphatase | 26 [NA to NA] — Measure of dispersion was not calculated for median change from baseline.

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Anidulafungin-Voriconazole
Serious Adverse Events (participants affected / at risk) | 29/54
Other Adverse Events (participants affected / at risk) | 26/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin-Voriconazole (N=54)
Blood disorder (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 4
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Pancreatic insufficiency (Gastrointestinal disorders) | 1
Death (General disorders) | 3
Drug ineffective (General disorders) | 1
Multi-organ disorder (General disorders) | 4
Pyrexia (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Abdominal sepsis (Infections and infestations) | 1
Abdominal wall abscess (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Fusarium infection (Infections and infestations) | 1
Pelvic infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia klebsiella (Infections and infestations) | 1
Pulmonary sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 11
Anastomotic leak (Injury, poisoning and procedural complications) | 1
Failure to anastomose (Injury, poisoning and procedural complications) | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Leukaemia recurrrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Partial seizures (Nervous system disorders) | 1
Anuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Arterial thrombosis (Vascular disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Hypovolaemic shock (Vascular disorders) | 1
Lupus vasculitis (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin-Voriconazole (N=54)
Anaemia (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Pyrexia (General disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
Protocol registration indicated timeframes for EIVT and/or Week 2 F/U for time to event, mortality, vital signs, and labs; however, analyses were continuous and reported from baseline to EIVT (up to Day 42), Week 2 F/U, or Week 6 telephone F/U visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.